CLINICAL TRIAL: NCT05185102
Title: Modeling Variation of the Objective Mental Workload for Tasks Requiring Different Cognitive Functions.
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Nantes University Hospital (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: RC21_0590
Record Dates: First submitted 2021-12-23; First posted 2022-01-11 (Actual); Last update posted 2022-09-27 (Actual); Status verified 2022-09

CONDITIONS: Healthy Subjects

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Cognitive tasks (Experimental): Electroencephalographic signals registration during different levels of difficulty of three tasks requiring very distinct cognitive functions: the updating of verbal memory, visuospatial span and mental motor inhibition.
  Interventions: Other: Cognitive tasks

INTERVENTIONS:
Other: Cognitive tasks — Electroencephalographic signals registration during different levels of difficulty of three tasks requiring very distinct cognitive functions: the updating of verbal memory, visuospatial span and mental motor inhibition.

SUMMARY:
This study focuses on the identification of objective mental workload (through ElectroEncephaloGraphy) during tasks involving different cognitive functions.

DETAILED DESCRIPTION:
In a medical context based on the solicitation of various cognitive functions, it is essential to be able to modulate the level of difficulty of the task, to maintain a constant level of mental workload while preserving the playful aspect of the activity. This must be sufficient to maintain the person's involvement without inducing too high a mental workload.

However, currently, there is no standardized model of variation of mental workload for cognitive tasks that could be used to modulate the difficulty. The present study is therefore part of this context and concerns the identification of the mental workload during tasks requiring cognitive functions such as memory or attention.

Further this study will allow to adapt in real time the difficulty of virtual tasks to the mental workload of people. In other words, to have a universal brain decoder of the mental workload.

ELIGIBILITY:
Inclusion Criteria:

* Age> 20 years old and <50 years old
* French-speaking men or women
* Fluent in French (native speaker or fluent)
* Hold at least a baccalaureate +2
* Right-handed
* Having normal or corrected to normal vision
* Having normal or corrected to normal hearing

Exclusion Criteria:

* Minors
* Adults under guardianship or curatorship
* Non-French speakers
* Sleep debt at the time of the experience
* Daltonism
* Vision and hearing uncorrected to normal
* Pregnant or breastfeeding women
* History of associated cranial trauma or any other neurological pathology altering the cerebral sensory-motor system or the cognitive capacities and higher functions.

Ages: 20 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 20 (Actual)
Dates: Start 2022-05-04 (Actual); Primary Completion 2022-06-23 (Actual); Study Completion 2022-06-23 (Actual)

PRIMARY OUTCOMES:
Identification of the variation in mental workload for different cognitive tasks. | Day 1
  Concomitant evolution in healthy volunteers of the ElectroEncephaloGraphic (EEG) signals and of the subjective mental workload for different levels of difficulty of three tasks requiring very distinct cognitive functions: the updating of verbal memory, visuospatial span and mental motor inhibition.

SECONDARY OUTCOMES:
Analysis of the influence of the quantity of EEG signals analyzed by our brain decoder on its accuracy | Day 1

CONTACTS AND LOCATIONS:
Overall Officials: Vincent ROUALDES, Doctor, Principal Investigator — Nantes University Hospital
Locations (1):
- Nantes University Hospital, Nantes, France

IPD SHARING:
Plan to Share IPD: No